CLINICAL TRIAL: NCT06657846
Title: Health-Related Quality of Life and Financial Toxicity in Patients With VEXAS Syndrome: An Italian GIMEMA Study
Brief Title: HRQoL and Financial Toxicity in Patients With VEXAS Syndrome
Status: Recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: QoL-Vexas
Record Dates: First submitted 2024-06-20; First posted 2024-10-26 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-10

CONDITIONS: VEXAS
MeSH Terms: conditions — VEXAS syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality of life assessment: Quality of life questionnaires

SUMMARY:
This multicenter cross-sectional observational study aims to describe health-related quality of life (HRQoL) and symptom profiles of patients with VEXAS syndrome.

DETAILED DESCRIPTION:
Moreover, the study will investigate financial toxicity and treatment tolerability. To contextualize the results the data of VEXAS patients will be compared with a cohort of matched MDS patients.

The overall aim of the study is to establish benchmark HRQoL data to be used in future prospective studies and clinical trial design.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) with a confirmed diagnosis of VEXAS syndrome (UBA1 pathogenic mutation detected)
* Written informed consent

Exclusion Criteria:

* - Having any kind of psychiatric disorder or major cognitive dysfunction.
* Not able to read and understand local language

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a confirmed diagnosis of VEXAS syndrome
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
EORTC QLQ-C30 | one time at study entry
  Mean score of EORTC QLQ-C30 scales (0-100):
  * 5 functional scales (physical, role, emotional, social, and cognitive)
  * global health status/QoL scale
    --> higher scores indicating better function, QoL
  * 3 symptom scales (fatigue, nausea and vomiting, pain)
  * 6 single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties)
    * higher scores indicating higher level of symptoms
FACIT-Fatigue | one time at study entry
  Mean score of FACIT-Fatigue (0 to 52)
  --> higher scores indicating higher levels of fatigue.

SECONDARY OUTCOMES:
PROFFIT-score | one time at study entry
  To investigate the association of the primary outcomes EORTC QLQ-C30, FACIT-Fatigue) and the PROFFIT-score (consisting of 7 items rated on a 4-point Likert scale)
Percentage of patients above previously validated cut-off scores for the EORTC QLQ-C30 indicating clinically relevant problems and symptoms | one time at study entry
  To assess the percentage of patients above previously validated cut-off scores for the EORTC QLQ-C30 indicating clinically relevant problems and symptoms
EORTC QLQ-C30 mean scale score stratified by age groups and sex. | one time at study entry
  To assess EORTC QLQ-C30 mean scale score stratified by age groups and sex.
  EORTC QLQ-C30 scales (0-100):
  * 5 functional scales (physical, role, emotional, social, and cognitive)
  * global health status/QoL scale
    * higher scores indicating better function, QoL
  * 3 symptom scales (fatigue, nausea and vomiting, pain)
  * 6 single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties)
    * higher scores indicating higher level of symptoms
FACIT-Fatigue mean score stratified by age groups and sex | one time at study entry
  To assess FACIT-Fatigue mean score stratified by age groups and sex. (0 to 52) --> higher scores indicating higher levels of fatigue.
Score of the FACIT item GP5 | one time at study entry
  To assess the score of the FACIT item GP5. Item GP5 from the FACIT Measurement System is a summary measure to assess the patient-reported overall impact of treatment toxicity on a 5-point Likert scale, with a higher score indicating higher treatment toxicity.
Compare EORTC QLQ-C30 mean scale scores with a matched case control group of MDS patients | one time at study entry
  To compare EORTC QLQ-C30 mean scales scores with a matched case control group of MDS patients.
  EORTC QLQ-C30 scales (0-100):
  * 5 functional scales (physical, role, emotional, social, and cognitive)
  * global health status/QoL scale
    --> higher scores indicating better function, QoL
  * 3 symptom scales (fatigue, nausea and vomiting, pain)
  * 6 single items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea, financial difficulties)
    * higher scores indicating higher level of symptoms
Compare FACIT-Fatigue mean score with a matched case control group of MDS patients | one time at study entry
  To compare FACIT-Fatigue mean score with a matched case control group of MDS patients (0 to 52) --> higher scores indicating higher levels of fatigue.

CONTACTS AND LOCATIONS:
Locations (17):
- Italy (17):
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona - Sod Clinica Ematologica, Ancona
  - Asst Papa Giovanni Xxiii - Ospedale Di Bergamo - Sc Ematologia, Bergamo
  - Aou Di Bologna - Policlinico S. Orsola-Malpighi - Uoc Ematologia, Bologna
  - Asst Degli Spedali Civili Di Brescia - Uo Ematologia, Brescia
  - Istituto Di Candiolo - Fondazione Del Piemonte Per L'Oncologia - Irccs - Centro Trapianti, Candiolo
  - Aou Careggi - Firenze - Sod Ematologia, Florence
  - Fondazione Irccs Ca' Granda, Ospedale Maggiore Policlinico - Milano - Ematologia - Padiglione Marcora, Milan
  - Irccs Ospedale S. Raffaele - Milano - Uo Oncoematologia, Milan
  - Aou Federico Ii - Napoli - Uoc Ematologia, Napoli
  - Aou Di Padova - Uo Ematologia, Padua
  - Fondazione Ircss Policlinico San Matteo - Pavia - Uo Ematologia, Pavia
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova, Irccs - Sc Ematologia, Reggio Emilia
  - Aou Policlinico Tor Vergata - Roma - Uoc Trapianto Cellule Staminali, Roma
  - Ististuto Clinico Humanitas - Rozzano - Uo Oncologia Medica Ed Ematologia, Rozzano
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Ospedale Mauriziano Umberto I - Torino - Scdu Ematologia, Torino
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona